CLINICAL TRIAL: NCT06823310
Title: Antibiofilm Activity of Directly Printed Orthodontic Clear Aligners With Incorporated Chitosan Nanoparticles (A Randomized Clinical Trial)
Brief Title: Antibiofilm Activity of Chitosan Nanoparticles Incorporated Into Clear Aligners
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Malak Akram Alhuwaizi, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1015425
Record Dates: First submitted 2025-02-02; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Malocclusion, Angle Class I
Keywords: Clear Aligners; Chitosan; Nanoparticles; 3D printing; Anti-biofilm
MeSH Terms: conditions — Malocclusion, Angle Class I

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Other): control directly printed orthodontic clear aligners without chitosan nanoparticles
  Interventions: Device: Control (Standard treatment)
- chitosan (Experimental): Directly printed orthodontic clear aligners with chitosan nanoparticles
  Interventions: Device: Chitosan

INTERVENTIONS:
Device: Control (Standard treatment) — Directly printed orthodontic clear aligner without any additions
  Arms: Control
Device: Chitosan — Adding chitosan nanoparticles to directly printed orthodontic clear aligners in vivo to enhance anti- microbial activity against streptococcus mutans.
  Arms: chitosan

SUMMARY:
The use of orthodontic appliances and equipment has dramatically increased over the past few decades, mainly due to improvements in materials and manufacturing processes that have paved the way for improved treatments .

The preference for aligner treatment and the increase in its prevalence can be attributed to patient demand for "invisible" treatments and the limitations of conventional fixed orthodontics . Direct 3D printing offers the possibility of creating highly precise clear aligners with soft edges, digitally designed and identically reproduced for an entire set of treatment aligners. These provide a better fit, higher efficacy, and reproducibility .

Clear aligner treatment demonstrated promising results in terms of controlling plaque index, gingival health, and the prevalence of white spot lesions. Nevertheless, grooves, ridges, microcracks, and abrasions on the aligner surface provide a prime environment for bacterial adherence and the development of plaque biofilms. Adding chitosan, a minimally toxic agent with antibacterial properties and the ability to reduce enamel demineralization, to 3D-printed aligner resin materials may decrease the incidence of WSLs . Currently, there is limited research on including nanoparticles in aligners' material for microbe inhibition and, to the best of our knowledge, none of the research has assessed and compared the effect of adding chitosan to an aligner's resin.

DETAILED DESCRIPTION:
The use of orthodontic appliances and equipment has dramatically increased over the past few decades, mainly due to improvements in materials and manufacturing processes that have paved the way for improved treatments .

The preference for aligner treatment and the increase in its prevalence can be attributed to patient demand for "invisible" treatments and the limitations of conventional fixed orthodontics. Direct 3D printing offers the possibility of creating highly precise clear aligners with soft edges, digitally designed and identically reproduced for an entire set of treatment aligners. These provide a better fit, higher efficacy, and reproducibility.

Clear aligner treatment demonstrated promising results in terms of controlling plaque index, gingival health, and the prevalence of white spot lesions. Nevertheless, grooves, ridges, microcracks, and abrasions on the aligner surface provide a prime environment for bacterial adherence and the development of plaque biofilms. A combination of mechanical and chemical methods seem to be a successful approach for removing plaque biofilm from aligners whilst preventing pigment adsorption.

Orthodontic appliances change the ecological environment of the oral cavity, resulting in a significant increase in the number of cariogenic bacteria such as Streptococcus mutans (S. mutans). The imbalance in oral homeostasis can lead to enamel demineralization, periodontitis and other bacteria-related adverse effects of orthodontic treatment. According to evidence-based clinical assessments, once enamel demineralization is formed it is difficult to be fully reversed using currently available remineralizing agents. Thus, several antibacterial strategies have been used clinically to prevent enamel demineralization, including antibacterial mouthwashes and toothpastes. However, these conventional interventions are largely dependent on perfect compliance from the patients, which most of the times does not occur.

Chitosan nanoparticles have a wide range of applications and have long been employed with or without other substances and techniques to increase their functionality .

Adding chitosan, a minimally toxic agent with antibacterial properties and the ability to reduce enamel demineralization, to 3D-printed aligner resin materials may decrease the incidence of WSLs . Currently, there is limited research on including nanoparticles in aligners' material for microbe inhibition and, to the best of our knowledge, none of the research has assessed and compared the effect of adding chitosan to an aligner's resin . A recent study carried out by Taher and Rasheed in 2023 added chitosan nanoparticles at different concentrations (2%, 3%, and 5% w/w) to directly 3D-printed clear aligner resin and assessed its anti-biofilm activity (on Streptococcus mutans bacteria categorized as one of the most virulent bacteria to cause enamel lesions), degree of conversion, accuracy, deflection force, and tensile strength. Additionally, cytotoxicity has been assessed using tissue cultures of mice fibroblasts and embryonic cells of chitosan (2%, 3%, and 5% w/w). The results of this essay showed that all used concentrations were non cytotoxic to living cells. It was found that there was a notable reduction in bacterial colonies when the resin was incorporated with 3% and 5% chitosan nanoparticles. No significant changes in the cytotoxicity or accuracy were detected and it was concluded that integrating biocompatible chitosan nanoparticles into the resin can add an anti-biofilm element to an aligner without compromising the material's particular biological, mechanical, and physical qualities at specific concentrations.

As the previous study was carried out in vitro, this study aims at assessing the effect of in vivo aging on the anti-biofilm and anti-microbial activity of chitosan incorporated into directly printed clear aligner resin.

ELIGIBILITY:
Inclusion Criteria:

* Subjects falling in the age group of 18-28 years with mild malocclusion
* Full permanent dentition except for third molars
* Plaque score and Bleeding on probing should be less than 10% (O'Leary et al., 1972)
* No previous history of para-functional habits

Exclusion Criteria:

any criteria not mentioned above

-

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-04-25 (Estimated); Study Completion 2025-05-25 (Estimated)

PRIMARY OUTCOMES:
Antimicrobial properties of chitosan nanoparticles incorporated into directly 3D printed clear orthodontic aligner will be assessed by using antibiofilm assay | 2 weeks
  The main outcome of this study is yo determine the antimicrobial effect of chitosan nanoparticles directly added to 3D printed clear aligners against Streptococcus mutans. This will be conducted by using antibiofilm activity test at baseline, 1 week, and 2 weeks following wearing conventional and chitosan-incorporated clear aligners. From each device retrieved from the patients at these timepoints, a 5mm diameter disc will be cut from the labial aspect of the devices. These discs will be cultured overnight in a broth containing equal number of S. mutans bacteria. After 24 h, the number of vital bacteria and the biomass will be measured to determine the antibiofilm activity of chitosan-incorporated devices vs control.

SECONDARY OUTCOMES:
Self-reported questionnaire about satisfaction of wearing clear aligner (control and experimental) | 2 weeks
  To asses perceived patients outcome i.e., degree of satisfaction by using a questionnaire designed for this purpose about wearing both devices (control and experimental). The questionnaire consists of two sections. The first section is dedicated for collecting demographic and lifestyle variables. The second section is designed to assess the degree of satisfaction by answering close-end questions. Each positive response will be scored as "1" while negative response will be scored "0". The sum of these responses will represent the overall satisfaction for each patient.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, University of Baghdad, Baghdad, Al-Resafa, Iraq

IPD SHARING:
Plan to Share IPD: No